CLINICAL TRIAL: NCT05156333
Title: Probiotics in Pregnancy and Rectovaginal Group B Streptococcus (GBS) Colonization
Brief Title: Probiotics and GBS Colonization in Pregnancy
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Uneffective
Sponsor: University of Modena and Reggio Emilia (Other)
Collaborators: Daniela Menichini (Unknown); Maria Longo (Unknown)
Responsible Party: Principal Investigator, Prof. Fabio Facchinetti, Director of the Obstetrics and Gynecolocy department, University of Modena and Reggio Emilia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AOU 0025949/19
Record Dates: First submitted 2021-10-05; First posted 2021-12-14 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: GBS Rectovaginal Colonization; Neonatal Sepsis
Keywords: Probiotics; Pregnancy; GBS colonization
MeSH Terms: conditions — Neonatal Sepsis | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Multicenter, prospective, randomized, placebo-controlled, double-blind, parallel-group study aimed at underestimating the feasibility and effect of the use of probiotic starting from week 30 on vaginal / rectal colonization of GBS in women at low obstetric risk.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The randomization (1: 1) will take place in each center, using the same allocation sequence, in blocks of 4, with the indication of the treatment code inserted in a white, closed envelope. The code will correspond to the number written on the packages to be administered and the list of codes containing the definition of the treatments, will be kept in a sealed envelope, by a collaborator of the PI (Head Nurse), and opened upon completion of the study or at the time of need, in case maternal-fetal or neonatal serious adverse event.
  No member of the research team knows which treatment the patients receive because both the active and the placebo are packaged identically and are contained in identical white boxes. Only the randomization numbers distinguish them.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Daily oral administration of 1 capusle of placebo, composed of: hydroxypropylmethylcellulose; Anti-caking agent: Magnesium salts of fatty acids, Dioxide of silicon; Dye: E171.
  Interventions: Dietary Supplement: Respecta
- Probiotic (Active Comparator): Daily oral administration of 1 capsule of mixture of probiotics and milk glycoproteins with prebiotic action); Cornstarch; Anti-caking agents: Vegetable magnesium stearate, Silicon dioxide; Capsule orally administered: Hydroxypropylmethylcellulose (coloring: E171).
  Interventions: Dietary Supplement: Respecta

INTERVENTIONS:
Dietary Supplement: Respecta — Respecta® complex (mixture of probiotics and milk glycoproteins with prebiotic action); Cornstarch; Anti-caking agents: Vegetable magnesium stearate, Silicon dioxide; Capsule orally administered: Hydroxypropylmethylcellulose (coloring: E171).
  Daily oral administration of two capsules of the Giellepi Spa class IIa medical device "Respecta" or placebo, to be taken with a glass of water preferably between meals, starting from the 30th week of pregnancy until the 37th week after having vagino-rectal swab screening performed.
  Other Names: Probiotic

SUMMARY:
Multicentric, randomized, placebo-controlled, double-blind, parallel group study aimed at evaluating the feasibility and effect of the use of probiotic starting from the 30th week, on vaginal / rectal colonization of GBS in women at low obstetric risk.

DETAILED DESCRIPTION:
Multicenter, randomized, placebo-controlled, double-blind, parallel group study aimed at evaluating the feasibility and effect of the use of probiotic starting from the 30th week, on vaginal / rectal colonization of GBS in women at low obstetric risk.

The study includes low obstetric risk pregnant women within the 33rd week of gestation, with vaginal delivery expected. It excludes women who during pregnancy had a positive urine culture for GBS, women with a previous newborn suffering from early sepsis, use of antibiotics in the month prior to enrollment, women unable to understand the study and sign informed consent.

Intervention Daily oral administration of two capsules of the Giellepi Spa class IIa medical device "Respecta" or placebo, to be taken with a glass of water preferably between meals, starting from the 30th week of pregnancy until the 37th week after having vagino-rectal swab screening performed.

ELIGIBILITY:
Inclusion Criteria:

* low obstetric risk pregnant women by the 33rd week of gestation,
* vaginal delivery expected.

Exclusion Criteria:

* positive urine culture for GBS,
* previous newborn suffering from early sepsis,
* use of antibiotics in the month prior to enrollment,
* women unable to understand the study and sign informed consent.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 402 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
GBS Rectovaginal colonization | at 35-37 weeks
  Rate of colonized GBS pregnant (carriers) at the time of antepartum screening (35-37 ^ week).

SECONDARY OUTCOMES:
Intrapartum antibiotics profilaxisi | during labor
  Rata of women requiring antibiotic profilaxis intrapartum

OTHER OUTCOMES:
PROM | pre-labor
  Prelabor rupture of membranes evaluated according to clinical signs or fibronectin test
Pathologic APGAR score | at delivery
  The Apgar score is a measure of a baby's condition after birth. It guides midwives, doctors and nurses as to whether a baby needs immediate treatment or monitoring. It is used to check a newborn baby born at 1 minute and 5 minutes after their birth. It is named after Dr Virginia Apgar who developed the score.
  The Apgar score goes from 0 to 10 and it is classified as pathologic when is </= 7
Need for neonatal antibiotics | within the first 48 hours after birth
  Rate of neonates requiring antibiotics within the first 48h of life
Neonatal sepsis | within the first week after birth
  Rate of neonates developing a sepsis

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Ospedale dei Bambini "Vittore Buzzi", Milan, MI
  - Arcispedale Santa Maria Nuova Reggio Emilia, Reggio Emilia, RE
  - University Hospital of Modena, Modena

IPD SHARING:
Plan to Share IPD: Undecided